CLINICAL TRIAL: NCT01469988
Title: The VO2 Increase With Testosterone Addition - Heart Failure (VITA-HF) Trial
Acronym: VITA-HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 82-VH-01
Record Dates: First submitted 2011-11-02; First posted 2011-11-10 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2014-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone (Experimental)
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator)
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Patients will be dosed accordingly: Female: 0.3g once daily (or matching placebo) gel;Males: 5g once daily (or matching placebo) gel.

SUMMARY:
Evaluate the efficacy and safety of testosterone supplementation on functional capacity, biomarkers, quality of life and clinical outcomes for patients with heart failure.

DETAILED DESCRIPTION:
Background:Heart failure is a prevalent condition of major public health importance that leads to significant morbidity and mortality despite the use of current evidence-based therapy. Further development of novel therapies to alleviate symptoms, improve functional status and ultimately clinical outcomes are needed. Cardiac function alone cannot explain all aspects of the heart failure syndrome: hence a search for peripheral mechanisms and inter-connected cardiac and non-cardiac pathways has ensued. Testosterone plays an integral role in multiple organ systems for growth, development and maintenance of health with known effects on peripheral musculature, vasculature, sympathetic tone, endothelial function and restoration of muscle metabolic function which would be beneficial in HF. Chronic HF has been associated with reduced testosterone levels, and low testosterone levels have been linked to reduced VO2, increased BNP and ANP levels, and worse clinical outcomes. Testosterone supplementation acts as a peripheral vasodilator and acutely increases cardiac output,which would improve oxygen delivery to skeletal muscles and secondarily delay transfer to anaerobic metabolism and depletion of high-energy phosphates. The increase in muscle mass associated with testosterone therapy may also result in increased endurance and decreased muscle fatigability in HF patients. Early small trials demonstrate safety, tolerability and an improvement in exercise walking distance in patients with HF. We contend that the time is now ripe for an adequately-powered phase II trial in order to test if this therapy can improve symptoms and functional status for patients with heart failure.

Specific Aim:Evaluate the efficacy and safety of testosterone supplementation on functional capacity, biomarkers, quality of life and clinical outcomes for patients with heart failure.

Synopsis:We propose a phase II randomized controlled, multi-center, double-blind trial, "The VO2Increase with Testosterone Addition - Heart Failure (VITA-HF) Trial". We plan to enroll 318 patients with chronic HF and NYHA II-III in a 1:1 trial of testosterone therapy (versus placebo): our primary objective is to test the effects on peak VO2 at 26 weeks (a commonly used surrogate outcome in phase II HFRCTthat represents both central and peripheral effects of our interventions). Given the assumptions made (a peak VO2 standard deviation of 2.7 mls/kg/min, paired t-test, and 2-sided alpha 0.05), 318 patients will have 85% power to detect a 1.0 ml/kg/min difference between the groups in the change in peak VO2 over 26 weeks. The minimally clinically important difference for peak VO2 may be as small as 0.26 mls/kg/min but is possibly higher and therefore, we have taken a conservative approach similar to that of other CIHR and NIH trials. Additional measures of quality of life, biomarkers (BNP) and clinical outcomes will be performed at 26 and 52 weeks. Quantitative measurement of core laboratory echocardiographic imaging will also assess the effect on left ventricular remodeling and markers of systolic and diastolic function. Assessment at 26 weeks will allow for the early effects to be demonstrated whereas our secondary endpoint evaluated at 52 weeks will demonstrate clinical and other outcomes important for phase III planning (including clinical, biochemical and echocardiographic endpoints).Androgel 5g was selected due to compliance and prior RCT dosing to ensure efficacy with a broad safety margin.

Feasibility:The investigators on this grant are attending physicians in large, tertiary care heart failure clinics with large patient populations and extensive experience with recruiting patients into clinical studies. The 7 sites selected have both experience and expertise in enrolling HF patients in CIHR and NIH trials.

Importance:Our proposed trial (VITA-HF) tests a novel strategic target which could enhance the quality and potentially the quantity of life of patients with heart failure by modulating complementary peripheral and central HF mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* NYHA Class II - III
* Left ventricular ejection fraction available by echo, nuclear or MRI < 12 months
* On optimal medical therapy (as per CCS guidelines for Chronic Heart Failure)42 for >3 months
* Female patients only: participants must be >1 year post-menopausal (defined as 12 months of spontaneous amenorrhea and confirmed by screening FSH >40 mIU/mL) OR >6 weeks post surgical bilateral oophorectomy if surgically sterilized.

Exclusion Criteria:

* Already or likely to receive LVAD or organ transplant within 6 months
* History of illicit drug use or alcohol abuse within <3 months, or history of HIV, Hepatitis B or C
* History of hypertrophic obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, clinically significant congenital heart disease, severe aortic or mitral regurgitation or stenosis
* Non-cardiovascular diagnosis with reduced life expectancy < 1 year including active cancer
* Recent (<1 month) cardiovascular event (admission to hospital for unstable angina, acute coronary syndrome, hypertensive crisis or ventricular arrhythmia) or cerebrovascular event (transient ischemic attack or stroke) or recent (<3 months) implantation of cardiac resynchronization therapy
* Hematocrit > 48%
* Male patients only: PSA > 4 ng/ml, or presence of a prostate nodule
* Total serum testosterone > 350 ng/dl (12.1 nmol/L)
* Untreated severe obstructive sleep apnea per American Thoracic Society criteria
* Chronic glucocorticoid, or anabolic steroid therapy
* Chronic hemodialysis, serum creatinine > 264 umol/L (3 mg/dL) or eGFR< 15 ml/min (MDRD)
* Participation in a competing trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
In patients with chronic heart failure, does 26 weeks of treatment with transdermal testosterone improve peak VO2? | 26 weeks
  The primary endpoint is change in peak VO2 measured at baseline and 26 weeks. The timing of the primary endpoint was chosen to allow for effects of either therapy to be seen within a reasonable timeframe, and to minimize loss to follow up, withdrawal due to clinical or adverse events and published data thus far supporting that an effect could be seen within 26 weeks.

SECONDARY OUTCOMES:
In patients with chronic heart failure, does 26 or 52 weeks of treatment with transdermal testosterone improve quality of life, biomarker (b-type natriuretic peptide, fasting glucose) or echocardiographic measures (LVEF, LVEDD, LVESD, SV)? | 52 weeks
  Includes total hospitalizations or ED visits (total, CV and HF), change in serum BNP at 26 and 52 weeks, change in quality of life assessed by KCCQ and FACIT-F, and changes in echocardiographic parameters (change from baseline in LVEDD, LVESD, LVEF, or SV). The FACIT-F was developed to assess fatigue, and has been validated and used in RCT. Markers of testosterone status will be evaluated to evaluate that the levels of these individual markers are attained relative to the doses used.
In patients with chronic heart failure, does 52 weeks of treatment with transdermal testosterone reduce ED visits or hospitalization for heart failure, or total mortality? | 52 weeks
  Incorporates clinical endpoints and quality of life to determine if patients are improved, unchanged or worsened at 52 weeks. All patients will be ranked sequentially into a ranking stratified to 3 tiers: (1) Death [time to death from randomization date with earliest death given lowest rank]; (2) Cardiovascular hospitalization or ED visit [time to hospitalization or ED visit from randomization date, if alive]; and (3) Change in KCCQ score [if alive and no hospitalization or ED visit, then patients with least change are ranked lowest, unchanged ranked next and improvement ranked highest].

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ezekowitz, Principal Investigator — University of Alberta
Locations (7):
- Canada (7):
  - Ajax / Pickering, Ajax
  - Brampton (McMaster University), Brampton
  - Foothills Hospital (University of Calgary), Calgary
  - The University of Alberta (Mazankowski Alberta Heart Institute):, Edmonton
  - Surrey Memorial Hospital (University of British Columbia), Surrey
  - Toronto General Hospital (University of Toronto):, Toronto
  - Vancouver General Hospital (University of British Columbia), Vancouver